CLINICAL TRIAL: NCT02436044
Title: Hepatic Arterial Infusion Chemotherapy Using Oxaliplatin Plus Fluorouracil/Leucovorin for Patients With Locally Advanced Hepatocellular Carcinoma
Brief Title: HAIC Using Oxaliplatin Plus Fluorouracil/Leucovorin for Patients With Locally Advanced HCC
Status: Approved for marketing | Type: Expanded Access
Sponsor: Ming Zhao (Other)
Responsible Party: Sponsor-Investigator, Ming Zhao, Chief physician in Minimally Invasive Interventional Division,Medical Imaging Center,Sun Yat-sen University Cancer Center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2015-FXY-011
Record Dates: First submitted 2015-05-03; First posted 2015-05-06 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma; Injury; Blood Vessel, Hepatic, Artery
Keywords: Hepatocellular Carcinoma; Locally advanced stge; HAIC; FOLFOX4; Locally advanced
MeSH Terms: conditions — Carcinoma, Hepatocellular; Wounds and Injuries | interventions — Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Procedure: HAIC using oxaliplatin plus fluorouracil/leucovorin — Hepatic arterial infusion chemotherapy using oxaliplatin plus fluorouracil/leucovorin
Drug: Oxaliplatin — Oxaliplatin, 130mg/m2, intraarterial infusion for 2 hours, on day 1,every 3 weeks
Drug: Fluorouracil — Fluorouracil, 1-st.400mg/m2, bolus injection, on day 1,every 3 weeks 2-nd.2400mg/m2, intraarterial infusion for 46 hours, on day 1-2,every 3 weeks
Drug: Leucovorin — Leucovorin, 200mg/m2, intraarterial infusion for 2 hours, on day 1,every 3 weeks

SUMMARY:
A large proportion of Asian patients with HCC present with locally advanced or metastatic disease,at which point they are ineligible for curative treatments.Oxaliplatin plus fluorouracil/leucovorin intravenous infusion was proved effective in prolonging progression-free survival(PFS) than doxorubicin as palliative chemotherapy in patients with advanced HCC from Asia. Besides, hepatic arterial infusion chemotherapy (HAIC）is a widely used method for primary or metastasis liver tumor with high local tumor response. To our knowledge, there have not been any prospective studies to assess the safety and effecacy of HAIC using oxaliplatin plus fluorouracil/leucovorin for patients with locally advanced HCC.Thus,the purpose of this phase 2 study was to assess the safety and effecacy of HAIC using oxaliplatin plus fluorouracil/leucovorin for patients with locally advanced HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common malignancy worldwide and much more common in male than in female. Each year, the number of patients with HCC in China alone contributes to about 50% of the total cases and deaths in the world. In men, poor prognosis makes HCC the second most frequent cause of cancer-related mortality in less developed countries. Locally advanced or metastatic disease is found in 60%-70% of HCC patients at the time diagnosed, with a median survival time of only 3-4 months due to unavailability of potentially curative therapies. Therefore, treatments that can control the progression and improve the prognosis of advanced HCC are under great need in sufficient liver reservation. Recently, an oral multi-tyrosine kinase inhibitor sorafenib, was reported to significantly prolong overall survival (OS) and delay disease progression in patients with advanced HCC. To date, sorafenib is still the only standard treatment for advanced HCC approved by FDA. However, low response rates, modest survival advantages, high-level heterogeneity of individual response and relatively high cost, such limitations of sorafenib prohibit its widespread use in advanced HCC and more alternative therapies are highly required at present.

In fact, for the past 30 years, researchers never stop searching for effective chemotherapeutic agents for HCC, and a wide spectrum of cytotoxic drugs have been reported by a variety of studies, including doxorubicin, gemcitabine, capecitabine, 5-fluorouracil (5-FU), cisplatin and so on. Unfortunately, low and heterogeneous responses and the well-known toxic effects caused by chemotherapy severely slowed down the pace of drug development for HCC. Until last year, based on a multicenter randomized clinical trial known as the EACH study, Qin et al. reported that FOLFOX4 (oxaliplatin [OXA], leucovorin [LV], 5-FU) regimen was associated with significant better OS than doxorubicin regimen (5.7 vs. 4.3 months; hazard ratio: 0.74; P = 0.03) in Chinese subgroup that accounted for 75% of the EACH study population. This study has provided proof to suggest that the FOLFOX4 regimen may become a potentially more efficacious alternative to doxorubicin in Chinese patients with advanced HCC.

However, systemic toxicity of chemotherapy and impaired liver function is still a concern that could not be neglected. Compared with systemic chemotherapy, hepatic arterial infusion chemotherapy (HAIC) can provide chemotherapeutic agents to liver at higher concentration with lower toxicity and has been reported favor results in patients with advanced HCC. Additionally, for patients who are not initially eligible for curative treatment, e.g., resection or liver transplantation, HAIC may down disease stage and offer them a chance to undergo such treatment which gives good long-term results. Though various agents such as 5-FU and cisplatin were studied with HAIC, by far, there have been no data about the use of more effective regimens FOLFOX4 in HAIC. Therefore, we carried out a multi-center, prospective trial to investigate the effect and safety of HAI combined with FOLFOX4 regimens in Chinese population with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* No extrahepatic spread on imaging, and filfill one of them as follows: 1.multiple HCC lesions,> 5.0 cm in diameter;2.Portal venous hepatic vein/tumor thrombus or arteriovenous/portal fistula;3.Direct invasion adjacent organs except gallbladder or penetrate the peritoneum;4.diffuse HCC.
* Eastern Cooperative Oncology Group Performance Status 0-2
* Child-Pugh Stage A or B
* At least one evaluable intrahepatic target lesions
* Previous accept sorafenib but stoped for more than 4 weeks because of disease progression or intolerance to sorafenib or refused to recieved sorafenib
* Stoped for more than 4 weeks after local treatments(surgical resection, radiofrequency ablation, transcatheter arterial chemoembolization) of tumor if presence
* Sign the informed consent.

Exclusion Criteria:

* Ever received oxaliplatin or fluorouracil/leucovorin;
* A platelet counts of > 60,000/mm3, prothrombin time activity <40%;
* Albumin <2.8 g/dL, total bilirubin ≥51.3 umol/L; alanine aminotransferase (ALT) and aspartate transaminase（AST）≥5 times of upper limit
* Uncontrolled or refractory ascites, ongoing variceal bleeding or encephalopathy;
* Severe heart, brain or kidney diseases
* Previous or concurrent cancer that is distinct in primary site or histology from HCC
* Pregnant women or lactating women;
* Allergy to fluorouracil, oxaliplatin, leucovorin calcium or iodine contrast agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Minimally Invasive Interventional Division, Medical Imaging Center, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu S, Lai J, Lyu N, Xie Q, Cao H, Chen D, He M, Zhang B, Zhao M. Effects of Antiviral Therapy on HBV Reactivation and Survival in Hepatocellular Carcinoma Patients Undergoing Hepatic Artery Infusion Chemotherapy. Front Oncol. 2021 Feb 1;10:582504. doi: 10.3389/fonc.2020.582504. eCollection 2020. PMID 33614477